CLINICAL TRIAL: NCT07396233
Title: Effects of Diagonal Proprioceptive Neuromuscular Facilitation Patterns on Pain and Functional Outcomes in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Rabia Hassan, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBC KU-549/2025
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthristis; Osteearthritis; Knee Pain Arthritis
Keywords: Knee Osteoarthritis; Functional Disability; Knee Pain; Conventional Training; Osteoarthritis; Arthritis; Musculoskeletal Disease; Joint Disease
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Musculoskeletal Diseases; Joint Diseases | interventions — Diathermy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analyst will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diagonal Proprioceptive Neuromuscular Facilitation (PNF) Pattern Exercises + Heat Therapy. (Experimental): This arm will receive PNF pattern exercises using Diagonal 1 and Diagonal 2 Lower Limb Patterns of PNF and the heat therapy
  Interventions: Other: Diagonal Proprioceptive Neuromuscular Facilitation (PNF) Pattern Exercises; Other: Heat Therapy
- Conventional Strength Training Exercises + Heat Therapy (Active Comparator): This arm will receive evidence based treatment of Quadripceps and Hip Abductor Strengthening exercises and the heat therapy.
  Interventions: Other: Conventional Strength Training Exercises; Other: Heat Therapy

INTERVENTIONS:
Other: Diagonal Proprioceptive Neuromuscular Facilitation (PNF) Pattern Exercises — Diagonal PNF pattern exercises include Diagonal 1 and Diagonal 2 lower limb pattern movements performed against resistance to improve strength, flexibility, and functional performance.
  Arms: Diagonal Proprioceptive Neuromuscular Facilitation (PNF) Pattern Exercises + Heat Therapy.
Other: Conventional Strength Training Exercises — The conventional strength training exercises include quadriceps and hip abductor strengthening performed using resisted active movements to improve muscle strength and functional ability.
  Arms: Conventional Strength Training Exercises + Heat Therapy
Other: Heat Therapy — Heat therapy will be given for 10 minutes by the help of electric heating pad.

SUMMARY:
A randomized controlled trial will be conducted at the Department of Physiotherapy, Dr. Ziauddin Hospital and Al-Rayaz Hospital, Karachi, Pakistan. A total of 150 patients diagnosed with knee osteoarthritis, aged between 40-60 years, will be recruited through a non-probability purposive sampling technique. Written informed consent will be obtained from all eligible participants prior to enrollment. The participants will be randomly allocated by the help of computer generated randomization sheet, into two groups i.e. experimental and the control group, with 75 participants in each group. Group A (experimental group) will receive diagonal proprioceptive neuromuscular facilitation (PNF) pattern exercises, while Group B (control group) will receive conventional strength training exercises. Heat therapy will be administered to both groups. All participants will be assessed using a standardized assessment form. Outcome measures will include pain intensity, knee range of motion, functional disability, hamstring flexibility, dynamic balance, and fatigue level. A single blinded assessor will assess all participants at baseline and at post intervention. Treatment sessions will be given thrice a week on alternate days for 6 weeks.

DETAILED DESCRIPTION:
The Statistical Package for the Social Sciences (SPSS) version 23 will be used for data analysis. Mean and standard deviation will be calculated for quantitative variables such as age. Qualitative variables will be presented as frequencies and percentages. Outcome measures (decrease pain intensity, improve functional disability, increase knee range of motion, improve hamstring flexibility, dynamic balance, and fatigue level) recorded at baseline and after 18th session of intervention will be compared and analyzed. Repeated measures ANOVA will be applied for statistical analysis. A p-value of less than 0.05 will be considered as the level of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Both male and females with an age range between 40-60 years.
* Patients diagnosed with unilateral or bilateral Knee OA.
* Grade-II or grade-III on kellgren and Lawrence classification.
* Patients having pain intensity more than 3.4 cm on VAS as minimum cut off value.
* Duration of knee OA more than 3 months (chronic).

Exclusion Criteria:

* Patients with any neurological disorder.
* History of lower limb arthroplasty or any other knee surgery.
* Septic knee arthritis.
* Inflammatory rheumatic disease such as rheumatoid arthritis and gout.
* Cancer or any other malignancy such as bone tumor.
* Knee deformities such as contracture, genu valgum and genu varum.
* History of ligamentous injury and meniscal tear.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-07 (Actual); Primary Completion 2027-01-19 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity will be assessed with Visual Analogue Scale | Baseline and after 6 weeks of intervention
  The Visual Analogue Scale is a unidimensional measure of pain intensity, used to record patients' pain progression, or assess pain severity in different conditions. It is 0 to 10 cm scale. Patients rate their pain on the scale. Higher the score in centimeter, severe will be the pain experienced.
Change in range of motion will be assessed with Universal Goniometer | Baseline and after 6 weeks of intervention.
  The universal goniometer is an instrument for the precise measurement of range of movement angles in degree, especially one used to measure the angles before and after range of motion. Increase in the degree of angle suggests increase in range of movement.

SECONDARY OUTCOMES:
Change in functional disability will be assessed with Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline and after 6 weeks of intervention.
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems regarding functional disability. It consists of total 100 scores. Increase in scores suggests better function and decrease in scores suggests increased functional disability.
Change in hamstring flexibility will be assessed with Active Knee Extension test. | Baseline and after 6 weeks of intervention.
  The Active Knee Extension (AKE) test will be used to assess hamstring muscle length using a goniometer with the hip flexion position at 90°. A greater knee extension angle indicates greater hamstring muscle length.
Change in dynamic balance will be assessed with Four Step Square Test (FSST) | Baseline and after 6 weeks of intervention.
  The Four Square Step Test will be used to assess dynamic balance. It is measured in seconds. A higher completion times indicate poorer dynamic balance and a greater risk of falls.
Change in fatigue level will be assessed with Multidimensional Fatigue Inventory questionnaire. | Baseline and after 6 weeks of intervention.
  The multidimensional fatigue inventory is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Higher total scores correspond with more acute levels of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Hassan, MSAPT, Principal Investigator — Ziauddin University; Basit Ansari, PhD, Study Chair — University of Karachi; Aftab Ahmed Mirza Baig, PhD, Study Director — IQRA University
Locations (2):
- Pakistan (2):
  - Al-Rayaz Hospital, Karachi, Sindh
  - Dr. Ziauddin Hospital, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No
Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators interested in physical medicine rehabilitation and knee osteoarthritis management.

REFERENCES:
- [Background] Nafees K, Baig AAM, Ali SS, Ishaque F. Dynamic soft tissue mobilization versus proprioceptive neuromuscular facilitation in reducing hamstring muscle tightness in patients with knee osteoarthritis: a randomized control trial. BMC Musculoskelet Disord. 2023 Jun 2;24(1):447. doi: 10.1186/s12891-023-06571-y. PMID 37268961
- [Background] Mondorf K, Kaufman DB, Carbonell RG. Screening of combinatorial peptide libraries: identification of ligands for affinity purification of proteins using a radiological approach. J Pept Res. 1998 Dec;52(6):526-36. doi: 10.1111/j.1399-3011.1998.tb01257.x. PMID 9924997
- [Background] Gallo R, Rivara G, Cattarini G, Cozzani E, Guarrera M. Allergic contact dermatitis from myrrh. Contact Dermatitis. 1999 Oct;41(4):230-1. doi: 10.1111/j.1600-0536.1999.tb06143.x. No abstract available. PMID 10515111
- [Background] Song Q, Shen P, Mao M, Sun W, Zhang C, Li L. Proprioceptive neuromuscular facilitation improves pain and descending mechanics among elderly with knee osteoarthritis. Scand J Med Sci Sports. 2020 Sep;30(9):1655-1663. doi: 10.1111/sms.13709. Epub 2020 Jun 1. PMID 32407583